CLINICAL TRIAL: NCT00031785
Title: A Phase III, Double-Blind, Randomized Study of the Effect of Megestrol Acetate on Weight and Health Related Quality of Life in Lung Cancer Patients Receiving Thoracic Radiation Therapy
Brief Title: Megestrol in Treating Patients Who Are Undergoing Radiation Therapy for Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: REBACDR0000069226; CCCWFU-98199; NCI-P02-0210
Record Dates: First submitted 2002-03-08; First posted 2003-08-06 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Anorexia; Cachexia; Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; limited stage small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; anorexia; cachexia
MeSH Terms: conditions — Anorexia; Cachexia; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Megestrol Acetate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: megestrol acetate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Megestrol helps improve appetite. It is not yet known if megestrol is effective in limiting weight loss in patients who are undergoing radiation therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of megestrol in limiting weight loss in patients who are undergoing radiation therapy for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of megestrol on weight in patients receiving radiotherapy for lung cancer.
* Determine the quality of life of patients treated with this drug.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to histology (non-small cell lung cancer vs small cell lung cancer), and type of treatment (radiotherapy vs radiotherapy and non-cisplatin-containing chemotherapy vs radiotherapy and cisplatin-containing chemotherapy). Patients are randomized to one of two treatment arms.

All patients undergo thoracic radiotherapy beginning on week 1 and continuing for a total of 5-7 weeks.

* Arm I: Patients receive oral megestrol once daily beginning within the first 3 days of radiotherapy and continuing until 12 weeks after the completion of radiotherapy.
* Arm II: Patients receive oral placebo once daily beginning within the first 3 days of radiotherapy and continuing until 12 weeks after the completion of radiotherapy.

In both arms, quality of life is assessed at baseline, at the completion of radiotherapy, and at 4, 8, 12, 16, and 20 weeks after the completion of radiotherapy.

Patients are followed at 4 and 8 weeks.

PROJECTED ACCRUAL: A total of 98 patients (49 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed lung cancer

  * Unresectable stage I-IIIB non-small cell lung cancer (NSCLC)
  * Resected stage I-IIIB NSCLC
  * Limited stage small cell lung cancer
* Planned radiotherapy with a total dose of at least 5,000 cGy in fraction sizes of no greater than 200 cGy each
* No distant metastases
* No significant ascites, pleural effusions, or edema that would inhibit oral food intake or invalidate weight determinations

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled hypertension
* No active thromboembolic disease
* No myocardial infarction within the past 3 months
* No prior congestive heart failure or thromboembolic events

Pulmonary:

* No prior pulmonary edema

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 3 years except curatively treated carcinoma in situ of the cervix or non-melanoma skin cancer
* No uncontrolled diabetes with glycosylated hemoglobin greater than 10%
* No Cushing's syndrome
* No dietary restrictions (e.g., salt, sugar, or lipid)
* No other serious medical or psychiatric illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Endocrine therapy

Endocrine therapy:

* At least 12 months since prior corticosteroids, estrogens, progestins, or other steroid hormone except as antiemetic prior to chemotherapy
* No concurrent corticosteroids, estrogens, progestins, or other steroid hormone except as antiemetic prior to chemotherapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to lung

Surgery:

* See Disease Characteristics
* More than 14 days since prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2002-09-11 (Actual); Study Completion 2002-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States